CLINICAL TRIAL: NCT04388943
Title: Biomedical Research Informatics Centre for Cardiovascular Sciences (The BRICCS Study)
Status: Recruiting | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 14022
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Physiological Measurements Patient reported questionnaire Blood sampling

SUMMARY:
This project will examine the diagnosis and prognosis of patients with cardiovascular disease in hospital in- and outpatients and compare their characteristics with normal controls from the community. The cardiovascular diseases studied include coronary artery disease, heart failure, heart attacks, valve disease, cardiac surgery, dysrhythmias, aneurysms, embolism, strokes, peripheral vascular disease and hypertension. Current methods for diagnosis and predicting outcome in patients are limited and may lack accuracy. This study will collect clinical details, and blood and urine samples from patients for analysis of proteins, chemicals and genetic biomarkers which will enable an examination of the pathological mechanisms involved in cardiovascular disease. The data will also be used to improve diagnosis and also improve prediction of outcome in patients (future clinical events such as death, further hospitalisation with cardiovascular disease and the effects of any therapy given to the patients). In this way, we can develop accurate ways of assessing a patient's condition and how it could be effectively managed. The study will last for 20 years.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients and inpatients with cardiovascular disease, of either gender
* Aged 18-90 years old
* Examples of conditions include: coronary artery disease, heart failure, heart attacks (myocardial infarction), valve disease, cardiac surgery, dysrhythmias (including atrial fibrillation), aneurysms, embolism, strokes, peripheral vascular disease, hypertension (and its complications, such as left ventricular hypertrophy) or those presenting with chest pain
* Healthy volunteers
* Aged 18-90 years old
* From the community without cardiovascular or other diseases

Exclusion Criteria:

* Any patient who is unable to give consent
* Any patient with non-cardiovascular comorbidity likely to cause death within 6 months
* Patients know to be infected with HIV, Hepatitis B or any other agent posing an infection risk from unfixed material

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited from secondary care, inpatient and outpatient departments.
Sampling Method: Non-Probability Sample
Enrollment: 9500 (Estimated)
Dates: Start 2010-06-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To improve understanding of disease mechanisms in cardiovascular disease | 20 Years
  The principal objective is to improve upon our understanding of disease mechanisms in cardiovascular disease, using plasma and urine proteins or chemicals and a patient's genetic makeup, which may impact on the diagnosis and assessment of prognosis of cardiovascular disease.

SECONDARY OUTCOMES:
To improve prediction of responses to different treatments, using blood proteins or chemicals and a patient's genetic makeup | 20 Years
  Secondary objectives include predicting response to different treatments (which would include drugs, devices) using blood proteins or chemicals and a patient's genetic makeup, after appropriate matching by propensity scoring. Plus, assessing whether biomarkers in stool or other tissue can discern the presence and severity of coronary artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh J Samani, Professor, Principal Investigator — NIHR Leicester Biomedical Research Centre
Locations (1):
- University Hospitals Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No